CLINICAL TRIAL: NCT01902108
Title: Randomized Double-blind Trial Comparing the Post-operative Analgesic Efficacy of Local Wound Infiltration With Bupivacaine Alone to Bupivacaine With Clonidine in Posterior Spine Surgeries
Brief Title: Added Value of Local Clonidine for Spine Postoperative Pain Control, in Addition to Bupivacaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Responsible Party: Principal Investigator, Dr Joseph Maarrawi, Assistant Professor : Researcher - Pain Specialist - Neurosurgeon, St Joseph University, Beirut, Lebanon
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLON-POBPC
Record Dates: First submitted 2013-07-07; First posted 2013-07-18 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Post-operative Pain
Keywords: clonidine; bupivacaine; post-operative pain; arthrodesis; discectomy; local infiltration
MeSH Terms: conditions — Pain, Postoperative; Ankylosis | interventions — Bupivacaine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clonidine (Experimental): Clonidine 150μg added to bupivacaine in a local infiltration before wound incision
  Interventions: Drug: Clonidine
- Bupivacaine (Active Comparator): Bupivacaine 0.25 % alone in the wound infiltration
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Local infiltration before wound incision with 20 ml of Bupivacaine 0.25 % alone
  Arms: Bupivacaine
Drug: Clonidine — Clonidine 150μg locally infiltrated with 20 ml of bupivacaine 0.25 % before wound incision
  Arms: Clonidine

SUMMARY:
The objective of this prospective randomized double-blind study is to evaluate the added analgesic value of clonidine to the conventional local bupivacaine wound infiltration in posterior spine surgery.

DETAILED DESCRIPTION:
Patients candidates to posterior spine surgery (Micro-discectomy, Lumbar laminectomy with or without fusion, cervical laminectomy) are asked to participate to this prospective study. After verification of inclusion and exclusion criteria, patients consenting to enter the study are randomly assigned to one of the following subgroups: 1-Pre-incisional wound infiltration with 20 mL of bupivacaine 0.25%. 2- Pre-incisional wound infiltration with 150 μg of clonidine with 20 mL of bupivacaine 0.25%. Demographic parameters, co-morbidities and other pre and per operative medical data are noted. In the post-operative period, patients received a standardized post-operative analgesic protocol (NSAI and paracetamol). Patients are asked to fill their pain diary using Visual Analog Scale (VAS) from day 0 till day 8 after surgery. Morphine rescue consumption is noted. Finally, the percentage of global subjective patient satisfaction regarding the post-operative wound pain is noted from 0 to 100.

ELIGIBILITY:
Inclusion Criteria:

* First (not recurrent) posterior spinal surgery at the operated site
* American Society of Anesthesiologists class I or II (operative risk)

Exclusion Criteria:

* Allergy to local anesthetics or to clonidine
* Pregnancy
* Raynaud's syndrome
* Thromboangiitis obliterans
* History of substance abuse
* Current treatment with corticosteroids

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Mean Area under curve | From the day of surgery till the 8th postoperative day (9 days and 8 nights=200h
  Pain is assessed on numeric rating scale (NRS) 8times/day during the first 3 days, 3times/day during the next 6days and one mean value during the night. The mean intensity of daily pain is obtained from the different values mentioned during day and night corrected by the duration covered by every value. It may vary from 0 to 10.

SECONDARY OUTCOMES:
Area under Curve (AUC) of pain | Calculated at Day 0-2, Day3-5, Day6-8 and all along the follow-up from Day0 till Day8
  The AUC during an interval (in days) is calculated by adding the different values of pain assessed during day and night multiplied by the duration (in hours) of sufferance from this amount of pain. The AUC during an interval is proportional to the mean intensity of pain suffered during the same interval. It is expressed in pain unit multiplied by hour
Daily rescue opiates consumption | From the day of surgery till the 3rd postoperative day
  The unit of rescue opiates consumption equals the administration of 5mg of morphine subcutaneously. The minimum interval between 2 rescue opiates consumption is 6 hours. Thus, the rescue opiates consumption may vary from 0 to 4/day.
Global subjective patient satisfaction of post-operative wound pain control | Assessed at the end of follow-up on Day 8
  It may vary from 0 that means a total dissatisfaction to 100% that means a complete satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Maarrawi, MD, PhD, Principal Investigator — Laboratory of neurosciences, Faculty of medicine, St Joseph University of Beirut
Locations (1):
- Hotel Dieu de france Hospital, Beirut, Lebanon

REFERENCES:
- [Derived] Abdel Hay J, Kobaiter-Maarrawi S, Tabet P, Moussa R, Rizk T, Nohra G, Okais N, Samaha E, Maarrawi J. Bupivacaine Field Block With Clonidine for Postoperative Pain Control in Posterior Spine Approaches: A Randomized Double-Blind Trial. Neurosurgery. 2018 Jun 1;82(6):790-798. doi: 10.1093/neuros/nyx313. PMID 28973650